CLINICAL TRIAL: NCT06164990
Title: Polyether Ketone Ketone (PEKK) Framework for Mandibular Implant-supported Complete Fixed Dental Prostheses With All-on-four Treatment Concept Clinical and Radiographic Study
Brief Title: (PEKK) Framework for Mandibular Implant-supported Complete Fixed Prostheses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatma mahanna (Other)
Responsible Party: Sponsor-Investigator, Fatma mahanna, lecturer of prosthodontics, Mansoura University
Organization: Mansoura University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A01100522
Record Dates: First submitted 2023-12-02; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Bone Loss; Peri-Implantitis
MeSH Terms: conditions — Bone Diseases, Metabolic; Peri-Implantitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEKK (Pekkton) framework (Experimental): PEKK (Pekkton) framework in mandibular implant-supported complete fixed dental prostheses with All-on-four treatment concept and evaluated regarding peri-implant tissue health
  Interventions: Other: PEKK framework

INTERVENTIONS:
Other: PEKK framework — PEKK (Pekkton) framework in mandibular implant-supported complete fixed dental prostheses with All-on-four treatment concept

SUMMARY:
This clinical study aims to evaluate the effect of using PEKK (Pekkton) framework in mandibular implant-supported complete fixed dental prostheses with All-on-four treatment concept on peri-implant tissues health

DETAILED DESCRIPTION:
The aim of this clinical study is to evaluate the effect of using PEKK (Pekkton) framework in mandibular implant-supported complete fixed dental prostheses with All-on-four treatment concept on peri-implant tissues health regarding the following parameters:

* Modified Plaque index
* Modified Gingival index
* Peri-implant probing pocket depth

Radiographic evaluation (periapical x-ray):

Marginal bone height changes

ELIGIBILITY:
Inclusion Criteria:

* Maxillary and mandibular alveolar ridges were covered with healthy, firm, relatively even thickness and even compressible mucosa and free from any signs of inflammation or flabbiness.
* Patients had completely edentulous maxillary and mandibular ridges with sufficient mandibular bone height not less than 15 mm in the interforaminal area and at least 12mm posteriorly
* All patients had sufficient inter-arch space
* All patients complained of insufficient retention and stability of their conventional mandibular dentures.
* All patients were of Angel's class I maxillo-mandibular relationship.

Exclusion Criteria:

* Patients with absolute contraindications for implant placement, such as active cancer and diseases of the immune system.
* Patients with metabolic diseases that are directly related to bone resorption, such as uncontrolled diabetes, osteoporosis, and hyperparathyroidism.
* Patients with general contraindications for surgical procedures, such as hematologic diseases, hepatic patients, patients with bleeding disorders, and serious problems with coagulation.
* Patients with a history of irradiation of the head and neck region or chemotherapy in the last 3 years were also excluded.
* Patients with relative contraindications such as a history of parafunctional habits (such as bruxism and clenching), smoking, alcoholism, and patients with any physical reasons that could affect follow-up.
* Patients with local contraindications for implant placement, such as localized bone defects.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
peri-implant tissues health (Clinical) | 1 year
  Modified gingival index
modified plaque index | 1 year
  peri-implant tissues health (Clinical)
peri-implant probing depth | 1 year
  Probing depth using plastic periodontal probe
Peri-implant radiographic evaluation | 1 year
  Marginal bone height changes using periapical radiograph

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, mansoura university, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No